CLINICAL TRIAL: NCT00375622
Title: Anti-Estrogen Therapy for Hereditary Hemorrhagic Telangiectasia A Double-Blind Placebo-Controlled Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3393
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: HHT; Epistaxis; Tamoxifen; Hemoglobin
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen

SUMMARY:
Hereditary hemorrhagic telangiectasia (HHT) is associated with recurrent epistaxis in 90% of cases. Good response to hormone treatment has been documented, although its use remains controversial. A double-blind placebo-controlled trial with estrogen treatment did not show any benefit over placebo. The aim of this study is to examine the efficacy of an antiestrogenic agent, TAMOXIFEN, in the treatment of HHT-associated epistaxis. The study will include up to 60 patients, over 18 years old.

DETAILED DESCRIPTION:
Patients with HHT-related epistaxis who will attend our center will randomly be assigned to 6 months of treatment with either Tab. tamoxifen 20 mg once daily or placebo. The group will included both men and women over the age of 18 years.

A detailed medical history will be taken at presentation. All patients will be examined by an otolaryngologist before and during the trial to assess the nasal condition and telangiectases and blood clots in the airway, nasal and oral cavity, and body skin. Blood will be collected for blood count and measurement of clotting time and liver function at onset of the trial and once monthly during treatment. Patients will be requested to complete a daily chart describing the course of their epistaxis, and female patients will be referred for gynecologic follow-up, including ultrasound. Evaluations will be conducted once a month throughout the treatment period.

The study was approved by the Ethics Committee of Rabin Medical Center. All patients will sign a consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from HHT with severe epistaxis
* Over 18 years old

Exclusion Criteria:

* Under 18 years old
* Pregnancy
* Treatment with anticoagulance
* Treatment with hormones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-02; Study Completion 2006-06

PRIMARY OUTCOMES:
Frequency of epistaxis.
Duration of epistaxis.
Hemoglobin level.

SECONDARY OUTCOMES:
Quality of life.
Nasal airway.

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Yaniv, MD, Study Chair — Rabin Medical Center, Clalit Health Services
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel